CLINICAL TRIAL: NCT05423496
Title: KidneyCare Immuno-optimization in Renal Allografts
Brief Title: KidneyCare Immuno-optimization in Renal Allografts (KIRA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision based on clinical utility considerations
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SN-C-00013
Record Dates: First submitted 2022-05-31; First posted 2022-06-21 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant; Immunosuppression; Allograft
Keywords: Calcineurin inhibitors; allograft loss and survival; Chronic immunosuppression; Steroid avoidance; Low-risk kidney transplant recipients; Acute rejection; KidneyCare; Immunological risk assessment; Cross-match testing; Donor-specific antibodies; Donor-derived cell-free DNA; AlloSue; AlloMap; iBox; Gene expression profiling; HistoMap assay; Immune optimization
MeSH Terms: interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Steroid Control Arm (Active Comparator): 133 patient undergoing KidneyCare Surveillance with Immune optimization at clinician discretion
  Interventions: Diagnostic Test: KidneyCare
- Steroid Immuno-optimization Arm (Experimental): 267 patient undergoing KidneyCare Surveillance with protocolized AlloSure-guided immuno-optimization of steroids/CNI
  Interventions: Diagnostic Test: KidneyCare; Drug: steroid
- Tacrolimus and mycophenolate mofetil (MMF) Control Arm (Active Comparator): 133 patient undergoing KidneyCare Surveillance with Immune optimization at clinician discretion
  Interventions: Diagnostic Test: KidneyCare
- MMF Immuno-optimization Arm (Experimental): 267 patient undergoing KidneyCare Surveillance with protocolized AlloSure-guided immuno-optimization of MMF/CNI
  Interventions: Diagnostic Test: KidneyCare; Drug: MMF

INTERVENTIONS:
Diagnostic Test: KidneyCare — Using KidneyCare platform as a tool to successfully augment immunosuppressant agents through regular surveillance allowing minimization of doses and number of agents.
Drug: steroid — optimization of steroids
  Arms: Steroid Immuno-optimization Arm
Drug: MMF — optimization of MMF
  Arms: MMF Immuno-optimization Arm

SUMMARY:
This is an unblinded, randomized, four-arm interventional research study enrolling patients who are undergoing kidney transplantation. The aim of the study is to determine whether patients at low risk of rejection can safely reduce the doses of their post-transplant immunosuppression medications using a combination of tests that include donor-specific antibodies (DSA), histology (looking at tissue from the donor graft), and donor-derived cell-free DNA (AlloSure). Eligible participants will be randomized in a 2:1 ratio into one of two immune-optimization (intervention) arms or the corresponding observational (control) arms. Two thirds of the participants in the study will have their decision to reduce immunosuppression made based on these test results and the other third will have the decision made based on standard of care clinical assessment and laboratory testing. The study will include two additional parameters under investigation - the AlloMap Kidney gene expression profiling test and the iBox prediction algorithm, but these will not be actively used to make any decisions as part of the trial. AlloSure, AlloMap Kidney, and iBox are the three components of the KidneyCare panel developed by CareDx.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label randomized controlled four-arm interventional trial of kidney transplant recipients receiving KidneyCare (AlloSure-Kidney, AlloMap Kidney, and iBox) surveillance testing. Eligible patients who meet inclusion/exclusion criteria and provide consent will undergo standard immune induction per their center protocol and begin a post-transplant maintenance regimen of tacrolimus and mycophenolate mofetil (MMF), with or without steroids after transplantation. If all prerequisite criteria are satisfied at 3 months, participants will be randomized and participants in the intervention arms will begin protocolized immuno-optimization, with the objective of the study being the gradual elimination of one immunosuppressive agent (either MMF or steroids) and optimization of calcineurin inhibitors (CNI) dosing. Any immune optimization changes in the control/observational arms will occur based on clinician discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the trial
2. Patients aged 18 years or older
3. cPRA <20% & no preformed DSA at time of transplant (using center-specific threshold)
4. Recipient (or planned recipient, if pre-transplant) of single, first-time, deceased (DBD/DCD) or living donor Kidney Transplant
5. Planned post-transplant maintenance immunosuppression regimen consisting of tacrolimus and MMF, with or without prednisone
6. Negative virtual crossmatch (performed by transplant center)
7. Female participants of childbearing potential must be willing to ensure that they or their partner use effective contraception during the trial
8. In the Investigator's opinion, is able and willing to comply with all trial requirements

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

1. Female participant who is pregnant, lactating, or planning pregnancy during the trial
2. Preformed DSA or ABO incompatible transplant
3. Chronic oral steroid use (for any reason)
4. Planned post-transplant immunosuppression regimen utilizing cyclosporine, azathioprine, mTOR inhibitors, and/or co-stimulatory blockers
5. Donor organ from identical twin or history of prior kidney transplant
6. Multivisceral transplant (heart/kidney, kidney/pancreas, liver/kidney, etc.) or history of hematopoietic stem cell transplant
7. Participant with life expectancy of less than 6 months or is inappropriate for immuno-optimization (including those patients at increased risk of primary disease recurrence w/ reduction in post-transplant immunosuppression)
8. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
9. Participants who are currently or have previously participated in another research trial involving an investigational drug/product in the past 12 weeks
10. Any condition that would preclude protocol biopsies (e.g. patients on lifelong anticoagulation for whom anticoagulation cannot be safely held)

Randomization Criteria (assessed at 3 months)

The participant may not proceed with randomization if ANY of the following apply:

1. Maintenance immunosuppression that includes cyclosporine, azathioprine, mTOR inhibitors, and/or co-stimulatory blockers
2. Baseline proteinuria ≥0.5g/day (confirmed by repeat measurement)
3. Baseline eGFR <45mL/min (average of 3 most recent prior readings)
4. Any episodes of biopsy-proven acute rejection (TCMR ≥1A or ABMR) since the time of transplant
5. Any interval detection of de novo DSA since the time of transplant (per center-specific threshold)
6. AlloSure result >0.5% at Month 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-02-23 (Estimated); Study Completion 2023-02-23 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) at 12 months, non-inferiority | 12 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (safety endpoint)
Estimated glomerular filtration rate (eGFR) at 24 months, non-inferiority | 24 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (safety endpoint)
Interstitial fibrosis/tubular atrophy (IF/TA) quantified by Banff Working Group biopsy grade(s) at 12-months post-transplant | 12 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (safety)
Interstitial fibrosis/tubular atrophy (IF/TA) quantified by Banff Working Group biopsy grade(s) at 24-months post-transplant | 24 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (safety)
Transplant glomerulopathy (TG) at 12-months post-transplant, quantified by biopsy-based histopathology grade(s) | 12 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (safety)
Transplant glomerulopathy (TG) at 24-months post-transplant, quantified by biopsy-based histopathology grade(s) | 24 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (safety)
Total number of biopsies performed post-transplant, including both surveillance and clinically indicated biopsies | 24 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (efficacy)
Number of clinically indicated biopsies planned and performed in the first 12- months post- transplant | 12 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (efficacy)
Number of clinically indicated biopsies planned and performed in the 24-months post- transplant | 24 months
  Demonstrate the safety and efficacy of KidneyCare as tool to successfully adjust immunosuppressant agents using regular surveillance for safe drug minimization. (efficacy)

SECONDARY OUTCOMES:
Histological assessment of tissue biopsy with paired AlloSure dd-cfDNA result - performed both 'For Cause' and 'Surveillance', using standard biopsy and HistoMap molecular assessment using nCounter. | 24 months
  Identify correlation between dd-cfDNA and histopathological allograft rejection based on all clinical biopsies.
Results of DSA testing, performed as outlined in the testing schedule | 24 months
  Compare rates of de-novo DSA antibody formation in immuno-optimization and control groups.

OTHER OUTCOMES:
Incidence of clinically-relevant infections among study participants (defined as infection requiring inpatient admission for evaluation/treatment) | 24 months
  Assessment of all medical events throughout the duration of the study.
Correlation between longitudinal AlloMap Kidney Scores / iBox Results and dosing of immunosuppressive agents | 24 months
  Assess utility of AlloMap Kidney and iBox results for purposes of immuno-optimization and post-transplant surveillance
Correlation between longitudinal AlloMap Kidney Scores / iBox Results and eFGR. | 24 months
  Assess utility of AlloMap Kidney and iBox results for purposes of immuno-optimization and post-transplant surveillance
Correlation between longitudinal AlloMap Kidney Scores / iBox Results and dnDSA rate. | 24 months
  Assess utility of AlloMap Kidney and iBox results for purposes of immuno-optimization and post-transplant surveillance
Correlation between cross-sectional AlloMap Kidney Scores / iBox Results and rejection (TCMR, ABMR) on histology from for-cause & surveillance biopsies. | 24 months
  Assess utility of AlloMap Kidney and iBox results for purposes of immuno-optimization and post-transplant surveillance
Correlation between cross-sectional AlloMap Kidney Scores / iBox Results and severity/grading of transplant glomerulopathy and IFTA on for-cause & surveillance biopsies | 24 months
  Assess utility of AlloMap Kidney and iBox results for purposes of immuno-optimization and post-transplant surveillance
Immunosuppression Dosing | 24 months
  Comparison of cumulative immunosuppression exposure in each arm (average daily dose over time)
Immunosuppression Exposure | 24 months
  Comparison of final dosage of each immunosuppressive agent at the conclusion of the study in each arm (tacrolimus, mycophenolate/Myfortic, prednisone)
Incidence of viremia ( including BK & CMV), defined as copies/mL in excess of the limit of detection | 24 months
  Assessment of all medical events throughout the duration of the study
PCR viral load over time (defined as time to resolution after initial identification of infection) | 24 months
  Assessment of all medical events throughout the duration of the study
Incidence of any associated end-organ manifestations of viral infection | 24 months
  Assessment of all medical events throughout the duration of the study
Changes in immunosuppression, defined as the change in the median daily dose (mg/day) of immunosuppressive agents | 24 months
  Assessment of all medical events throughout the duration of the study
Incidence of proteinuria, defined by urine protein to creatinine ratio >0.5g/g, confirmed on serial samples | 24 months
  Assessment of all medical events throughout the duration of the study
Number of clinically defined and/or biopsy-confirmed allograft rejection events, including the specific histologic diagnosis made, and if treated, description and duration of therapeutic regimen | 24 months
  Assessment of all medical events throughout the duration of the study